CLINICAL TRIAL: NCT03569696
Title: Improving the Outcome of High-risk Aggressive B-cell Lymphoma Patients With Nivolumab Maintenance Therapy. The NivoM Trial
Brief Title: Improving the Outcome of High-risk Aggressive B-cell Lymphoma Patients With Nivolumab Maintenance Therapy
Acronym: NivoM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meirav Kedmi MD (Other Government)
Responsible Party: Sponsor-Investigator, Meirav Kedmi MD, Dr. Meirav Kedmi, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-18-4728-MK-CTIL
Record Dates: First submitted 2018-06-13; First posted 2018-06-26 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Lymphoma, B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Single Group Assignment All the participating patients will receive 240mg nivolumab every 2 weeks for 8 doses for 4 months, and later 480 mg every 4 weeks for 2 years (cycle 9-30) for a maximum of 30 doses, starting 10±2 weeks after the last cycle of immunochemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Nivolumab will be administered intravenously every 2 weeks in a dose of 240mg over 30 minutes for 8 cycles and then 480mg every 4 weeks for two years (cycle 9-30)to a maximum of 30 doses whichever comes first.
  Interventions: Biological: nivolumab

INTERVENTIONS:
Biological: nivolumab — The treatment phase will begin 10 ± 2 weeks from completion of R- anthracycline based therapy. Cycle 1 day 1 will occur within 72 hours from enrolment. Study treatment will be continued until nivolumab discontinuation due to disease progression, unacceptable toxicity or completion of 2 years or 30 doses of therapy. Study drug nivolumab will be administered intravenously every 2 weeks as described in the investigator brochure (IB) in a dose of 240mg over 30 minutes 46 for 8 cycles and then 480mg every 4 weeks for two years (cycle 9-30)to a maximum of 30 doses whichever comes first.

SUMMARY:
This trial is designed as a unicenter, single arm phase II trial. The aim of the trial is to test whether prognosis of high-risk Aggressive B cell Lymphoma (ABCL) patients who are in complete remission (CR) post immunochemotherapy can be improved by 2year nivolumab maintenance therapy. Participants will be recruited from Chaim Sheba Medical Center as well as from other medical centers in Israel through the Israeli lymphoma group. Therapy will be treated in Chaim Sheba Medical Center.

DETAILED DESCRIPTION:
The rationale for prolonged nivolumab therapy in high-risk ABCL patients in CR following 1st line standard therapy is based on the hypothesis that the stimulation of immune system by Programmed cell death protein 1 (PD1) blockade will also facilitate the eradication of minimal residual disease (MRD), that is not apparent by positron emission tomography (PET) imaging, and eventually will prevent relapse and improve survival. The Study will include adult patients, age ≥18, with high risk (IPI≥3) ABCL, in CR according to PETCT, as defined by the Lugano Criteria, following first-line rituximab (R) and anthracycline-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients age ≥18.
2. Histologically confirmed DLBCL, primary mediastinal B cell lymphoma or any other aggressive B-cell lymphoma as defined by the World Health Organization (WHO) 2016 criteria 4, with IPI of 3 or more post completion R- anthracycline containing regimen for at least 6 cycles and in complete remission according to the Lugano Criteria 45 per PETCT.
3. Hematology laboratory values must be within the following limits:

   1. Absolute neutrophil count (ANC) ≥ 1000/mm3 independent of growth factor support
   2. Platelets ≥100,000/mm3 independent of transfusion support.
4. Biochemical values within the following limits:

   1. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x upper limit of normal (ULN)
   2. Total bilirubin ≤ 1.5 x ULN unless the increase is due to Gilbert's syndrome or of non- hepatic origin
   3. Serum creatinine ≤ 2 x ULN or estimated Glomerular Filtration Rate (Cockroft-Gault)

      * 40 mL/min/1.73m2
5. Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for 1 month after the last dose of study drug. For males, these restrictions apply for 3 months after the last dose of study drug.
6. Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [Beta-hCG]) or urine pregnancy test at screening. Women who are pregnant or breastfeeding are ineligible for this study.
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
8. Sign (or their legally acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study.

Exclusion Criteria:

1. Patients not in CR, as defined by the Lugano Criteria, after completion of first line R- anthracycline based therapy.
2. Patients previously treated with any line of therapy for relapsed/refractory disease.
3. Major surgery within 4 weeks of starting the first nivolumab infusion.
4. Previous treatment with nivolumab or any other PD-1 or PD-L1/2 inhibitors.
5. Prior allogeneic stem cell transplantation.
6. Known central nervous system lymphoma.
7. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
8. Clinically significant pulmonary disease.
9. Vaccinated with live, attenuated vaccines within 4 weeks of enrolment.
10. Known history of human immunodeficiency virus (HIV).
11. Active Hepatitis C Virus or active Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics. Hepatitis B core antigen (HBC) positive as well as HBs positive, HBcore positive HBs negative patients will not be eligible.
12. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety.
13. Patients with an active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
14. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
15. Diagnosed or treated for a malignancy other than DLBCL, except:

    1. Malignancy treated with curative intent and with no active disease present for 3 years before enrolment
    2. Adequately treated non-melanoma skin cancer or lentigo malignant without evidence of disease.
    3. Adequately treated carcinoma in situ without evidence of disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10-08 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
disease progression | 3 years post diagnosis of aggressive B cell lymphoma.
  To evaluate the proportion of high-risk ABCL patients with no evidence of disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Meirav Kedmi, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical organization, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No